CLINICAL TRIAL: NCT03678285
Title: Hematological Risk Factors Related to Acute Renal Injury During High Intensity Training
Brief Title: Acute Renal Injury During High Intensity Training
Acronym: HIFRT-KH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20180607EJ02013
Record Dates: First submitted 2018-08-30; First posted 2018-09-19 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Acute Kidney Injury; Exercise
Keywords: High intensity exercise; Proenkephalin-A
MeSH Terms: conditions — Acute Kidney Injury; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will take part in the same, single bout, exercise intervention
Masking Description: No other parties besides the participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFRT Workout (Experimental): Consecutive completion of; 1 mile run, 100 pull ups, 200 push-ups, 300 bodyweight squats, 1 mile run.
  Interventions: Other: HIFRT Workout

INTERVENTIONS:
Other: HIFRT Workout — A single high intensity functional resistance training (HIFRT) exercise bout.

SUMMARY:
The proposed work is designed to be the first in a series of studies investigating the health benefits and risks related to high intensity training (HIT) exercise. Our specific aims are to determine, 1) if participation in a single bout of HIT induces hematological markers consistent with acute kidney injury (AKI), and 2) if risk is predicted by the pre-exercise concentration of plasma proenkephalin-A.

This investigation is an observational case control study. In year one, data collection procedures will be refined with ~40 participants local to the University of Wyoming and training will occur for collaborators from Wyoming community and tribal colleges. In year two, data collection will expand to some of the 12 CrossFit® gyms in Wyoming with assistance from the community and tribal colleges. Blood and urine samples will be collected before and up to 48 h after a standardized bout of HIT exercise on ~100 participants. Baseline blood samples will be analyzed for proenkephalin-A. All blood samples will be analyzed for markers of muscle damage (e.g., creatine kinase and myoglobin), and markers of kidney function (e.g., serum creatinine and blood urea nitrogen). Urine will be analyzed for markers of filtration function (e.g., albumin, creatinine, neutrophil gelatinase-associated lipocalin [NGAL], and kidney injury molecule 1 [KIM-1]). Lastly, the severity of kidney damage will be compared with the number of risk alleles and proenkephalin-A concentration.

The investigators envision that the bout of HIT exercise will induce markers consistent with skeletal muscle damage in most participants and, based on literature from other styles of intense exercise, that acute kidney injury will be diagnosable in between 50-75% of participants. Secondarily, the investigators predict that the concentration of proenkephalin-A will be inversely related to the change in kidney function from before to after the HIT exercise bout.

DETAILED DESCRIPTION:
The HIT-KH investigation is proposed to take place over the course of two calendar years. During year one collaborations with gyms specializing in High Intensity Resistance and Functional Training style workouts (referred to from this point forward as satellite data collection sites) as well as community and tribal colleges (referred to from this point forward as partner institutions) local to these facilities will be solidified. Also, during the summer of year one data collection will occur on a small subset of individuals (~40) at a data collection site local to the University of Wyoming (Figure 1.). It is our plan to use this first data collection in Laramie, WY as a training session for all students from partner institutions so that the students are prepared when the data collection is expanded to the satellite data collection sites in year 2.

In order to properly power this investigation the investigators have estimated that about 100 participants will be needed. Given that the investigators can expect about 40 participants from the local Larmie data collection gym (CrossFit® 7220)this will require the investigators to partner with other high intensity resistance and functional training gyms around the state of Wyoming in year 2. The investigators have chosen to reach out to CrossFit® gyms specifically because it is common practice for most CrossFit® gyms to program the workout the investigators are interested in observing (Murph), at least once per year. Collection data on 60 additional participants will require partnership with 3 additional gyms (i.e., 20 participants / facility). At this point the investigators have been in contact with 3 gym owners all of whom have offered verbal agreement to assisting with data collection. Among these gyms is CrossFit® Leveler, located on the Wind River Reservation in Fort Washikie, Wyoming. This facility is a Native American owned business and it primarily caters to those Native American's living on the reservation. Because the state of Wyoming is ~2% Native American in population, the inclusion of this facility in our investigation is very important for proper sampling (see attached letter of support from owner Mike Ute). Additional gyms that have been contacted and are in the process of providing written approval are CrossFit® Frontier (Cheyenne), and, Cloud Peak CrossFit® (Sheridan).

Because our data collection will be occurring throughout the state the investigators also plan to partner with local community and tribal colleges local to many of the above satellite data collection sites. Briefly, the investigators plan to incorporate up to three students and one faculty mentor from each of the following educational institutions; Laramie County Community College, Wind River Tribal College, and Sheridan Community College. Regarding the inclusion of Wind River Tribal College and the Wind River Indian Reservation, Investigator Johnson is under the guidance of Dr. Christine Porter who is also in the University of Wyoming Division of Kinesiology and Health. Dr. Porter has successfully implemented several research studies on the Wind River Reservation and is well versed in the intricacies and requirements necessary for the completion of data collection in this partnership. Lastly, the partner institutions are beneficial to the project because the data collection takes place over the course of 5 consecutive days, training and working with local researchers will enable this project to reduce the cost because a large research team from Laramie, Wyoming will not be required for each data collection.

As mentioned above 1-3 students from each of the above institutions will be requested to assist with data collection for HIT-KH. Part of our grant funding is devoted to payment of fees for these student's training. This includes travel fees to travel and stay in Laramie, Wyoming during year 1 for observation and basic level assistance with the initial data collection. During the end of year 1 and/or beginning of year 2 additional funds have been allocated to provide phlebotomy training to interested students. These students will then be utilized during year two data collections to assist with blood draws. Finally, funds have been allocated for travel to and attendance of the Rocky Mountain Regional American College of Sports Medicine conference. It is our goal that at least one student will be able to use the preliminary data from the year 1 data collection to compile a research abstract that will be submitted for presentation. All other students will be offered the ability to attend and participate in the conference during the spring of 2019.

Blood samples will be collected one day before participants take part in the workout, and 24 and 48hrs after completion. Sampling will take place by single venipuncture to an antecubital vein by a trained investigator using sterile technique and universal precautions. Following any needle removal, firm pressure will be applied over the site of the blood draw with gauze to minimize the occurrence of a hematoma. Blood will be drawn into vacutainers specific for each of the analytes to be analyzed later. Tubes will be centrifuged as soon as possible, then the blood plasma, serum, or white blood cells will be removed and aliquoted into separate cryovials. These cryovials will be frozen in the -80C freezer as soon as possible. For satellite data collections, if -80C freezers are not available at the local partner institution, liquid nitrogen will be used to freeze and store samples until the samples can be transported back to the University of Wyoming for more permanent storage.

Urine samples will be collected in 24 hr collection jugs for the period immediately prior to the workout and for two 24hr periods following. Each sample will be weighed for measurement of total volume, evaluated for urine color and urine specific gravity. Dipsticks will be used on fresh samples while three 2mL aliquots of each 24hr sample will be separated and stored at room temperature until the samples are returned to the University of Wyoming where the samples will be frozen at -80C for future analysis.

Fresh 24hr urine samples will be analyzed using traditional dipsticks for the following variables: leukocytes, nitrite, urobilinogen, protein, pH, hemoglobin, ketone, bilirubin, and glucose. Additionally, fresh samples will be evaluated for urine color and specific gravity via handheld refractometer in order to establish hydration state. Further biochemical urinary analysis are reviewed below.

Proenkephalin-A will be analyzed at the Clinical Research Center by the use of a chemiluminometric sandwich immunoassay. The laboratory group in Malmo has previously successfully measured this hormone (Schulz et al., 2017). All remaining blood and urine samples will be analyzed within the Human Integrated Physiology laboratory located at the University of Wyoming using colorimetric enzyme-linked immunosorbent assays (ELISA). These samples will be analyzed for the following variables; serum creatinine, blood urea nitrogen, urinary creatinine, neutrophil gelatinase-associated lipocalin [NGAL], and kidney injury molecule 1 [KIM-1]). All ELISA antibodies will be supplied by "Abcam", (Cambridge, Massachusetts, USA) and microplates will be read according the manufacturer's instructions on spectrophotometer (Epoch 2, Biotek, Winooski, Vermont, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individual who has completed this specific workout on at least one prior occasion

Exclusion Criteria:

1. Score of "0" on the Functional Movement Screening (FMS) test as evaluated by two investigators * indicating pain during any of the seven functional movements
2. Self- reported Kidney (chronic kidney disease, polycystic kidney disease, glomerulonephritis, diabetic nephropathy, interstitial nephritis, Goodpasture syndrome) or other medical condition contraindicating participation in HIFRT (Hypertension, dyslipidemia, type II diabetes mellitus, BMI >30)
3. Pregnancy, suspected pregnancy, or breastfeeding
4. Blood donations within the last eight weeks leading up to testing day
5. Any musculoskeletal injuries which have resulted in > 1 week of absence from HIFRT within the last six months
6. Not passing the physical activity readiness questionnaire (PAR-Q)
7. Allergy to ibuprofen or non-steroidal anti-inflammatory medication
8. Surgical operation on digestive tract or kidneys, except appendectomy
9. Inability to participate in the entire study
10. Recurrent urinary tract infections or kidney stones
11. History of protein or blood in urine
12. Moving from a location of low altitude (< 3,000') to Laramie within the past 3 months
13. Inability to understand and write English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan C Johnson, PhD, Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poston WS, Haddock CK, Heinrich KM, Jahnke SA, Jitnarin N, Batchelor DB. Is High-Intensity Functional Training (HIFT)/CrossFit Safe for Military Fitness Training? Mil Med. 2016 Jul;181(7):627-37. doi: 10.7205/MILMED-D-15-00273. PMID 27391615
- [Background] Bergeron MF, Nindl BC, Deuster PA, Baumgartner N, Kane SF, Kraemer WJ, Sexauer LR, Thompson WR, O'Connor FG. Consortium for Health and Military Performance and American College of Sports Medicine consensus paper on extreme conditioning programs in military personnel. Curr Sports Med Rep. 2011 Nov-Dec;10(6):383-9. doi: 10.1249/JSR.0b013e318237bf8a. PMID 22071400
- [Background] Mansour SG, Verma G, Pata RW, Martin TG, Perazella MA, Parikh CR. Kidney Injury and Repair Biomarkers in Marathon Runners. Am J Kidney Dis. 2017 Aug;70(2):252-261. doi: 10.1053/j.ajkd.2017.01.045. Epub 2017 Mar 28. PMID 28363731
- [Background] Schulz CA, Christensson A, Ericson U, Almgren P, Hindy G, Nilsson PM, Struck J, Bergmann A, Melander O, Orho-Melander M. High Level of Fasting Plasma Proenkephalin-A Predicts Deterioration of Kidney Function and Incidence of CKD. J Am Soc Nephrol. 2017 Jan;28(1):291-303. doi: 10.1681/ASN.2015101177. Epub 2016 Jul 8. PMID 27401687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited between October 2018 and May 2019
Period: Overall Study
Arm/Group | HIFRT Workout
Started | 42
Started Workout | 40
Completed | 38
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by subject prior to start of workout | 1
Not completed — Dehydrated prior to start of workout | 1

BASELINE CHARACTERISTICS:
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 42
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — (mmHg). Taken at rest after sitting for 5 min with feet flat on ground. Measurements were repeated at 1 min interval until 2 measurements were within 2mmHg. Population: 4 participants discontinued participation after enrolling but prior to baseline measurements
  mmHg
    number analyzed (Participants) | 38
    (all) | 119 (11)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 4 subjects ended participation after enrollment but prior to baseline measurements.
  mmHg
    number analyzed (Participants) | 38
    (all) | 74 (7)
Visual Analog Pain Perception [Mean (Standard Deviation); unit: units on a scale] — Scale minimum = 0mm Scale maximum = 100mm
  0 is associated with the anchor "No Pain", 100 is associated with the anchor "Worst Possible Pain" Population: 4 subjects stopped participation after enrollment but prior to baseline measurements.
  units on a scale
    number analyzed (Participants) | 38
    (all) | 3 (6)
urinary neutrophil gelatinase-associated Lipocalin [Mean (Standard Deviation); unit: (ng/ml)/(ml/min)] — Population: 4 subjects stopped participation prior to baseline measurements. 2 subjects did not provide adequate baseline urine sample for analysis.
  (ng/ml)/(ml/min)
    number analyzed (Participants) | 36
    (all) | 9.2 (25.7)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — Population: 4 subjects stopped participation prior to baseline measurements
  mg/dL
    number analyzed (Participants) | 38
    (all) | 1.05 (0.16)
Proenkephalin [Mean (Standard Deviation); unit: pmol/L] — Population: 4 subjects stopped participation prior to baseline measurements
  pmol/L
    number analyzed (Participants) | 38
    (all) | 61.1 (16.9)
urinary kidney injury molecule 1 [Mean (Standard Deviation); unit: pg/mL] — Population: 4 subjects stopped participation prior to baseline measurements. 2 subjects did not provide adequate baseline urine samples for analysis.
  pg/mL
    number analyzed (Participants) | 36
    (all) | 170.5 (180.8)
Creatine Kinase [Mean (Standard Deviation); unit: U/L] — Population: 4 subjects stopped participation prior to baseline measurements. 1 participant sample was not available.
  U/L
    number analyzed (Participants) | 37
    (all) | 267.8 (185.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Concentration of Proenkephalin-A From Baseline to 4 Time-points Surrounding the Workout
Description: an endogenous opioid polypeptide hormone which, via proteolytic cleavage, produces the enkephalin peptides [Met]enkephalin, and to a lesser extent, [Leu]enkephalin.
Time Frame: Baseline, Immediately pre-exercise, immediately post-exercise, 24 hours post-exercise, 48 hours post-exercise
Population: Number analyzed for 48 hour post-exercise change is 1 less than total sample due to a blood sample that was not able to be analyzed at the final time point
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 38
pmol/L
  Immediately pre-exercise | 1.65 (13.18)
  Immediately post-exercise | 3.69 (15.49)
  24 hours post-exercise | 2.50 (12.58)
  48 hours post-exercise: number analyzed (Participants) | 37
  48 hours post-exercise | 2.13 (12.68)

2. Primary Outcome: Change in Serum Creatinine
Description: Marker of kidney function measured as a change in concentration between baseline to 4 time-points surrounding the workout
Time Frame: Baseline, Immediately pre-exercise, immediately post-exercise, 24 hours post-exercise, 48 hours post-exercise.
Population: One sample at the final time point was not able to be analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 38
mg/dL
  Immediately pre-exercise | 0.001 (0.066)
  Immediately post-exercise | 0.211 (0.119)
  24 hours post-exercise | 0.008 (0.062)
  48 hours post-exercise: number analyzed (Participants) | 37
  48 hours post-exercise | -0.014 (0.086)

3. Primary Outcome: Change in Creatinine Kinase
Description: Marker of skeletal muscle damage measured as a change in concentration between baseline and 4 time-points surrounding exercise
Time Frame: Baseline, Immediately pre-exercise, immediately post-exercise, 24 hours post-exercise, 48 hours post-exercise
Population: There is a discrepancy in the number of participants analyzed because one participant's samples were unable to be analyzed at all time points. One additional participant had a sample that was missing at the final time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 38
U/L
  Immediately pre-exercise | -48 (76)
  Immediately post-exercise | 98 (107)
  24 hours post-exercise | 781 (1631)
  48 hours post-exercise: number analyzed (Participants) | 36
  48 hours post-exercise | 1152 (2406)

4. Primary Outcome: Change in 24 Hour Urinary Kidney Injury Molecule 1
Description: Marker of Kidney Injury measured as a change in concentration between baseline to 2 time points surrounding exercise
Time Frame: Baseline, Day 2, Day 3
Population: One subject declined to collect 24hr urine at any time during the study. One subject did not provide an adequate sample for the baseline measurement (therefore no change scores could be calculated from baseline at either of the follow up points). Two additional subjects did not return complete collections on the final day of measurement
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 36
pg/mL
  Day 1 to Day 2 Change | 71.17 (132.63)
  Day 1 to Day 3 Change: number analyzed (Participants) | 34
  Day 1 to Day 3 Change | 45.44 (226.49)

5. Primary Outcome: Change in 24 Hour Urinary Neutrophil Gelatinase-associated Lipocalin
Description: Marker of kidney damage measured as a change in concentration between baseline and 2 time points surrounding the exercise
Time Frame: Baseline, Day 2, Day 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (ng/ml)/(ml/min)
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 36
(ng/ml)/(ml/min)
  Day 1 to Day 2 Change | 5.52 (20.94)
  Day 1 to Day 3 Change: number analyzed (Participants) | 34
  Day 1 to Day 3 Change | 2.50 (15.06)

6. Secondary Outcome: Change in the Short-form McGill Pain Questionnaire
Description: Subjective perception of muscle pain. The participant responds to 15 word prompts designed to describe types of pain (e.g., "shooting"), with "none", "mild", "moderate", or "severe". These are scored as 0, 1, 2, and 3 respectively. A participant's Pain Score is the cumulative score for all prompt responses added together. As a participant's total score increases this denotes greater subjective feeling of pain which may be associated with the above markers of skeletal muscle and/or kidney damage. The minimum score for this questionnaire is 0 and the maximum score is 45. Typically, the total score is only reported. However, if there are prompts (i.e., subscales) that are consistently rated high or low, we will report these as a way to further describe the type of pain that is being reported (e.g., "throbbing" versus "sharp"). This will only be done after the total score is reported.
Time Frame: Baseline, immediately pre-exercise, immediately post-exercise, 24 hours post-exercise, 48 hours post-exercise
Measure: Mean (Standard Deviation); unit: score on a scale in millimeters
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 38
score on a scale in millimeters
  Change to Immediately pre-exercise | -1 (5)
  Change to immediately post-exercise | 23 (23)
  Change to 24 hours post-exercise | 18 (16)
  Change to 48 hours post-exercise | 18 (17)

7. Secondary Outcome: Post Exercise Hypotension
Description: Systolic and Diastolic blood pressure measurements
Time Frame: Baseline, immediately pre-exercise, immediately post-exercise, 24 hours post-exercise, 48 hours post-exercise
Population: No blood pressure measurement was recorded for a single subject at the immediately pre-exercise time point.
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | HIFRT Workout
Number analyzed (Participants) | 38
mm/Hg
  systolic change to immediately pre-exercise: number analyzed (Participants) | 37
  systolic change to immediately pre-exercise | 3 (8)
  systolic change to immediately post-exercise | -8 (11)
  systolic change to 24 hours post-exercise | -3 (7)
  systolic change to 48 hours post exercise | -3 (8)
  diastolic change to immediately pre-exercise: number analyzed (Participants) | 37
  diastolic change to immediately pre-exercise | 2 (6)
  diastolic change to immediately post-exercise | -3 (6)
  diastolic change to 24 hours post-exercise | -3 (6)
  diastolic change to 48 hours post-exercise | -2 (5)

ADVERSE EVENTS:
Time Frame: During entire protocol enrollment. This was approximately 4 days (96 hours). Participants were able to contact investigators after 96 hours should they have experienced an adverse event following their final visit to the laboratory (i.e., allergy to bandage, increasing muscle soreness, etc.).
Arm/Group | HIFRT Workout
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 2/42
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIFRT Workout (N=42)
Ankle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 Participant strained ankle joint during the initial run portion of the workout and discontinued the workout at that point.
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 Participant experienced cramps in their quadriceps muscles during the squat portion of the workout. Their participation was terminated by investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03678285/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03678285/SAP_001.pdf